CLINICAL TRIAL: NCT07237230
Title: Clinical Study Protocol to Evaluate the Safety and Efficacy of γδ T Cells for the Prevention of Relapse After Allogeneic Transplantation in Patients With High-risk Acute Myeloid Leukemia
Brief Title: Clinical Study to Evaluate the Safety and Efficacy of γδ T Cells for the Prevention of Relapse After Allogeneic Transplantation in Patients With High-risk Acute Myeloid Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Donghua Zhang (Other)
Responsible Party: Sponsor-Investigator, Donghua Zhang, Director, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHZ1962-C
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: High-Risk Acute Myeloid Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Biological: allogeneic γδ T cell infusion

INTERVENTIONS:
Biological: allogeneic γδ T cell infusion — allogeneic γδ T cell infusion

SUMMARY:
This is an investigator-initiated clinical trial evaluating the safety and efficacy of allogeneic γδ T cell infusion for relapse prevention in high-risk acute myeloid leukemia patients after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signs the informed consent form and is expected to be able to complete the follow-up examinations and treatments required by the study procedures.
2. Age 18 to 65 years (inclusive), regardless of gender.
3. Patients have one of the high-risk factors for relapse before allogeneic hematopoietic stem cell transplantation：①Meets the diagnostic criteria for relapsed or refractory disease as defined by the Chinese Guidelines for Diagnosis and Management of Relapsed/Refractory Acute Myeloid Leukemia (2017 Edition);②Hyperleukocytosis (≥100×10⁹/L) with concomitant central nervous system leukemia (CNSL); ③Positive minimal residual disease (MRD) before transplantation; ④Populations defined as having poor prognosis;⑤Myelodysplastic syndromes transformed to or secondary acute myeloid leukemia.
4. Confirmed diagnosis of Acute Myeloid Leukemia(AML) and within 30±5 days after allogeneic transplantation.
5. The subject has recovered from toxicities of previous therapies, defined as CTCAE grade <2 (unless the abnormality is tumor-related or judged by the investigator to be stable with minimal impact on safety or efficacy).
6. Eastern Cooperative Oncology Group(ECOG) performance status score of 0-3 and an estimated life expectancy greater than 3 months.
7. Adequate organ function is defined as:

   1. Alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN);
   2. Aspartate aminotransferase (AST) ≤3 × ULN;
   3. Total bilirubin ≤1.5 × ULN;
   4. Serum creatinine ≤1.5 × ULN, or creatinine clearance ≥60 mL/min;
   5. Hemoglobin ≥50g/L (must not have received transfusion support within 7 days prior to laboratory testing);
   6. Room air oxygen saturation ≥92%;
   7. Left ventricular ejection fraction (LVEF) ≥45%, confirmed by echocardiography without pericardial effusion and no clinically significant ECG findings;
   8. No clinically significant pleural effusion.

Exclusion Criteria:

1. Diagnosis of another malignancy within 3 years prior to screening, except for adequately treated carcinoma in situ of the cervix, papillary thyroid carcinoma, basal cell or squamous cell skin cancer, localized prostate cancer after radical surgery, or ductal carcinoma in situ after radical surgery;
2. History of severe allergy (defined as a grade 2 or higher allergic reaction manifested by any of the following: airway obstruction [rhinorrhea, cough, wheezing, dyspnea], tachycardia, hypotension, arrhythmia, gastrointestinal symptoms [nausea, vomiting], incontinence, laryngeal edema, bronchospasm, cyanosis, shock, respiratory or cardiac arrest) or known allergy to any active ingredient, excipient, murine-derived products, or xenogeneic proteins contained in the investigational product;
3. Severe cardiac disease, including but not limited to severe arrhythmia, unstable angina, large-area myocardial infarction, New York Heart Association Class III or IV cardiac dysfunction, or refractory hypertension (defined as failure to achieve blood pressure control after >1 month of treatment with ≥3 tolerable antihypertensive drugs at optimal doses, including diuretics, or requiring ≥4 antihypertensive drugs for effective control);
4. Severe respiratory disease (including history of or concurrent severe interstitial lung disease, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, or symptomatic bronchospasm);
5. Presence of grade III-IV acute GVHD(Graft-Versus-Host Disease) or extensive chronic GVHD;
6. Current use (or intention to use) other maintenance therapies post-hematopoietic stem cell transplantation that have been demonstrated to adversely affect the persistence of γδ T cells in vivo;
7. Active neurological autoimmune or inflammatory diseases (e.g., Guillain-Barré syndrome [GBS], amyotrophic lateral sclerosis [ALS]) or clinically significant active cerebrovascular disease (e.g., cerebral edema, posterior reversible encephalopathy syndrome [PRES]);
8. Presence of severe psychiatric disorders;
9. History of alcohol abuse or drug abuse;
10. Clinically significant active cerebrovascular disease (e.g., cerebral edema, posterior reversible encephalopathy syndrome [PRES]);
11. Participation in another clinical study within 1 month prior to screening, unless deemed by the investigator as non-interfering with the safety and efficacy evaluation of the investigational product (e.g., non-interventional observational studies);
12. Women who are pregnant or breastfeeding, female subjects planning pregnancy within 1 year after cell infusion, or male subjects with partners planning pregnancy within 1 year after cell infusion;
13. Patients with contraindications to any study procedure or other medical conditions that may pose unacceptable risks, as determined by the investigator's judgment and/or clinical standards.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival (RFS) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China